CLINICAL TRIAL: NCT04609761
Title: Intravenous Immunoglobulin (IVIG) Treatment in Children With Pediatric Acute-onset Neuropsychiatric Syndrome (PANS): an Open-label Trial in South-western Sweden
Brief Title: Open-label Trial of IVIG in Children With PANS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IVIGPANSOpen
Record Dates: First submitted 2020-10-05; First posted 2020-10-30 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: PANS Pediatric Acute-Onset Neuropsychiatric Syndrome
MeSH Terms: conditions — Pediatric acute-onset neuropsychiatric syndrome | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Intervention Model Description: Open-label single-arm trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IVIG treatment (Experimental): Single-arm open-label
  Interventions: Drug: Privigen Injectable Product (Intravenous Immunoglobulin)

INTERVENTIONS:
Drug: Privigen Injectable Product (Intravenous Immunoglobulin) — Privigen, 2 g/kg BW every 4th week for 6 months (= 6 infusions).
  Other Names: IVIG

SUMMARY:
Open-label prospective trial to study efficacy, safety and tolerability of intravenous immunoglobulin (IVIG) once monthly for 6 months in children and adolescents with PANS. Number of subjects: 10. Age range: 4-17 years.

Pediatric Acute-onset Neuropsychiatric Syndrome (PANS) is a recently defined research diagnosis describing an abrupt, dramatic onset of neuropsychiatric symptoms including obsessions/compulsions and/or food restriction in children. Immunologic mechanisms are suspected, but treatment trials are few.

DETAILED DESCRIPTION:
Open-label prospective trial to study efficacy, safety and tolerability of intravenous immunoglobulin (IVIG) once monthly for 6 months in children and adolescents with PANS (including the subgroup PANDAS). Number of subjects: 10. Age range: 4-17 years.

Pediatric Acute-onset Neuropsychiatric Syndrome (PANS) is a recently defined research diagnosis describing an abrupt, dramatic onset of neuropsychiatric symptoms including obsessions/compulsions and/or food restriction in children. Immunologic mechanisms are suspected, but treatment trials are few.

The primary objective of this study is to evaluate the efficacy of intravenous immunoglobulin (IVIG), 2 g/kg given every 4 weeks for 6 months, to patients with post-infectious PANS/PANDAS, in improving neuropsychiatric symptoms and impairment.

The secondary objectives of this study are to evaluate changes from baseline to follow-up at 3 months, 6 months and 12 months in:

* Obsessive Compulsive Disorder (OCD) symptoms
* adaptive functioning
* quality of life
* cognitive functioning
* for patients with baseline inflammation signs on cerebral Magnetic Resonance Imaging (MRI) to evaluate changes in these measures after IVIG therapy after 6 months.
* number of days of work/school/daily activities missed per subject year due to PANS/PANDAS before and after IVIG therapy
* parental care load, e.g. need for sick leave, before and after IVIG therapy
* Immunoglobulin (IgG, IgM and IgA) levels at baseline, 3 months, 6 months and 12 months
* sustainability of any improvement at 12 months after initiation of IVIG measured with the PANS scale, CGI-S and CGI-I

To assess the safety and tolerability of high dose IVIG therapy

* Clinical signs and symptoms (nausea, headache, local reactions)
* ALAT
* Hemoglobin, complete blood count including leucocyte differential

Investigational product: Intravenous immunoglobulin IVIG (Privigen), 2 g/kg BW every 4th week for 6 months (= 6 infusions).

ELIGIBILITY:
Inclusion Criteria:

1. The subject and parents/caregivers have given written consent or assent to participate in the study.
2. Children and adolescents between the ages of 4 and 17 years at Baseline.
3. Documented and confirmed pre-existing diagnosis of post-infectious PANS/PANDAS
4. The subject has not been treated with IVIG previously or not been treated for the last 6 months
5. If the patient is on long-term antibiotic prophylaxis, this should be unchanged one month before baseline and during the trial. Throat culture for Group A Streptococcus (GAS) should be performed before study start and standard phenoxymethyl penicillin treatment given if positive culture.
6. Infections occurring during the trial should be treated according to standard clinical practice.
7. Treatment with COX-inhibitors or corticosteroids should be discontinued at least one month before baseline and during the trial. Two-three days treatment with corticosteroids during and after IVIG treatment is allowed to reduce IVIG side effects such as headache and nausea.
8. Any psychopharmacological treatment (e.g. SSRI, antipsychotics), if considered essential for the subject, should be kept at a stable and unchanged dose from one month before baseline and during the trial. If not considered essential, it should be discontinued at least one month before baseline.
9. The medical records for all subjects should be available to document diagnosis, previous infections and treatment.
10. For female participants, adequate contraception should be used, see exclusion criteria. A negative pregnancy test can possibly be a requirement, specify requirement/type of pregnancy test. Contraceptive requirements may also apply to male participants.

Exclusion Criteria:

1. Clinical evidence of any significant acute or chronic disease that, in the opinion of the Investigator, may interfere with successful completion of the trial or place the subject at undue medical risk. If encephalitis cannot be excluded by clinical history alone, spinal tap results are required before study start to rule out encephalitis (which would need to be treated according to encephalitis treatment guidelines). MRI should have been performed if clinically indicated.
2. The subject has had a known serious adverse reaction to immunoglobulin or any severe anaphylactic reaction to blood or any blood-derived product
3. Females of childbearing potential who are pregnant, have a positive pregnancy test at Baseline (human chorionic gonadotropin [HCG]-based assay), are breastfeeding, or unwilling to practice a highly effective method of contraception (oral, injectable or implanted hormonal methods of contraception, placement of an intrauterine device [IUD] or intrauterine system [IUS], condom or occlusive cap with spermicidal foam/gel/film/cream/suppository, male sterilization, or true abstinence) throughout the study Note: True abstinence: When this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods], declaration of abstinence for the duration of a trial, and withdrawal are not acceptable methods of contraception.)
4. The subject has significant proteinuria (dipstick proteinuria ≥ 3+, known urinary protein loss > 1 g/24 hours, or nephrotic syndrome), has a history of acute renal failure, has severe renal impairment (blood urea nitrogen [BUN] or creatinine more than 2.5 times the upper limit of normal [ULN]), and/or is on dialysis
5. The subject has Screening Visit values of aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels exceeding 2.5 times the ULN for the expected normal range for the testing laboratory.
6. The subject has hemoglobin < 90 g/L at Screening
7. The subject has a known previous infection with or clinical signs and symptoms consistent with current hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
8. The subject has a history of or current diagnosis of deep venous thrombosis or thromboembolism (e.g., myocardial infarction, cerebrovascular accident, or transient ischemic attack); history refers to an incident in the year prior to Baseline or 2 episodes over lifetime.
9. The subject currently has a known hyperviscosity syndrome
10. The subject has an acquired medical condition that is known to cause secondary immune deficiency, such as chronic lymphocytic leukemia, lymphoma, multiple myeloma, chronic or recurrent neutropenia (absolute neutrophil count less than 1.0 x 109/L], or HIV infection/acquired immune deficiency syndrome (AIDS).
11. The subject is HIV positive by NAT based on a Screening blood sample.
12. The subject has non-controlled arterial hypertension at a level of greater than or equal to the 90th percentile blood pressure (either systolic or diastolic) for their age and height
13. The subject is receiving any of the following medications: (a) immunosuppressants including chemotherapeutic agents, (b) immunomodulators, (c) long-term systemic corticosteroids defined as daily dose > 1 mg of prednisone equivalent/kg/day for > 30 days. Note: Intermittent courses of corticosteroids of not more than 10 days would not exclude a subject. Inhaled or topical corticosteroids are allowed.
14. The subject has known substance or prescription drug abuse.
15. The subject has participated in another clinical trial within 30 days prior to Baseline (observational studies without investigative treatments [non-interventional] are permitted) or has received any investigational blood product within the previous 3 months
16. The subject/caregiver is unwilling to comply with any aspect of the protocol, including IV infusions, blood sampling
17. Mentally challenged subjects who cannot give independent informed consent In the opinion of the Investigator the subject may have compliance problems with the protocol and the procedures of the protocol.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pediatric Acute-onset Neuropsychiatric Syndrome (PANS) scale symptoms and impairment | 6 months
  Investigator-rated scale measuring symptom severity and impairment in Pediatric Acute-onset Neuropsychiatric Syndrome (PANS), score range 0-50, lower is better
Change in CGI-S | 6 months
  CGI-S (Clinical Global Impression-Severity) measures global symptom severity, score range 1-7, lower is better
CGI-I | 6 months
  CGI-I (Clinical Global Impression-Improvement) measures global improvement, score range 1-7, lower is better

SECONDARY OUTCOMES:
Change in CY-BOCS scale | 6 months
  CY-BOCS scale measures Obsessive Compulsive Disorder (OCD) Symptoms, investigator-rated, score range 0-40, lower is better
Change on ABAS (Adaptive Behavior Assessment System) II scale | 6 months
  Measures level of functioning in everyday life, parent- and teacher-rated, score range 40-160, higher is better
Change on Child Health Inventory (CHIP-CE) scale | 6 months
  Measures quality of life, parent-rated, standardized T-score, mean 50, standard deviation 10, higher score is better
Change on 5-15 scale | 6 months
  Measures neuropsychiatric symptoms, score range 1-543, lower is better
Change in neuromotor functioning | 6 months
  Neuromotor examination by investigator
Change in cognitive function | 6 months
  Working memory test from Wechsler scale, standardized scores age norms, mean 100, standard deviation 10, higher is better
Change in School-PANS (Pediatric Acute-onset Neuropsychiatric Syndrome) Scale | 6 months
  Short version of PANS-scale rated by teacher or school assistant, score range 0-50, lower is better
School absence | 6 months
  Days absent from school past 3 months or since last visit
Parental care load | 6 months
  Sick leave number of days
Change in laboratory assessments | 6 months
  Inflammatory measures as specified in CRF, lower is better
Adverse events | 6 months
  Parent/child report
Magnetic Resonance Imaging (MRI) | 6 months
  In a subgroup who can tolerate MRI without general anaesthesia. Specially developed protocol for measuring inflammation signs

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Gillberg, Professor, Principal Investigator — Gillberg Neuropsychiatry, Centre Sahlgrenska Academy
Locations (1):
- Gillberg Neuropsychiatry Centre, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hajjari P, Oldmark MH, Fernell E, Jakobsson K, Vinsa I, Thorsson M, Monemi M, Stenlund L, Fasth A, Furuhjelm C, Johnels JA, Gillberg C, Johnson M. Paediatric Acute-onset Neuropsychiatric Syndrome (PANS) and intravenous immunoglobulin (IVIG): comprehensive open-label trial in ten children. BMC Psychiatry. 2022 Aug 6;22(1):535. doi: 10.1186/s12888-022-04181-x. PMID 35933358

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-29): https://cdn.clinicaltrials.gov/large-docs/61/NCT04609761/Prot_SAP_002.pdf